CLINICAL TRIAL: NCT03992716
Title: Reaching Protein Target With SmofKabiven® Extra Nitrogen Versus Olimel N9E: A Prospective, Randomised, Active-controlled, Patient-blinded, Multicentre Clinical Trial During the Early Phase of Acute Critical Illness
Brief Title: Reaching Protein Target With SmofKabiven® Extra Nitrogen vs Olimel N9E During the Early Phase of Acute Critical Illness
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study had to be put on hold after the outbreak of Covid-19 in the participating countries and was terminated in September 2020 since a date for re-starting was not foreseeable.
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SKNt-001-CP4; 2017-001972-46 (EudraCT Number)
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmofKabiven® extra Nitrogen (Experimental): Parenteral nutrition with SmofKabiven® extra Nitrogen in a dosage to provide 10 kcal/kg/day on Study Day 2 and 20 kcal/kg/day on Study Days 3 through 6.
  Interventions: Drug: SmofKabiven® extra Nitrogen
- Olimel N9E (Active Comparator): Parenteral nutrition with Olimel N9E in a dosage to provide 10 kcal/kg/day on Study Day 2 and 20 kcal/kg/day on Study Days 3 through 6.
  Interventions: Drug: Olimel N9E

INTERVENTIONS:
Drug: SmofKabiven® extra Nitrogen — SmofKabiven® extra Nitrogen (Fresenius Kabi) is a sterile, hypertonic emulsion for parenteral nutrition, in a 3-chamber bag containing amino acids, glucose, a lipid emulsion, and electrolytes.
  Arms: SmofKabiven® extra Nitrogen
Drug: Olimel N9E — Olimel N9E (Baxter) is a sterile, hypertonic emulsion for parenteral nutrition, in a 3-chamber bag containing amino acids, glucose, a lipid emulsion, and electrolytes.
  Arms: Olimel N9E

SUMMARY:
The main focus of the study is to show that SmofKabiven® extra Nitrogen, in a realistic clinical setting, enables to meet high protein requirements in patients during the first week after onset of critical illness, without risk of overfeeding with energy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <90 years, male and female
2. Critically ill, medical or surgical ICU patient
3. Admitted to the ICU on the same day or the day before with a minimum expected ICU stay of 3 days
4. Central venous access available for continuous infusion of the study drugs
5. Sequential Organ Failure Assessment (SOFA) score ≥2
6. Contraindication against enteral nutrition or limited tolerance to enteral nutrition and it is planned that patient receives ≥80% of the total target caloric intake from parenteral nutrition during the first 3 nutritional treatment days
7. Written informed consent from the patient or the patient's legal representative or deferred written consent from the patient or patient's legal representative (deferred proxy consent)

Exclusion Criteria:

1. Contraindication against parenteral nutrition or inability to receive parenteral nutrition via central venous access
2. Received parenteral nutrition within 7 days before randomisation
3. It is planned that patient receives ≥20% of the total target caloric intake via enteral or oral nutrition and/or non-nutritional sources (glucose solution for drug dilution or lipids from propofol/clevidipine or citrate from continuous renal replacement therapy) during the first 3 nutritional treatment days
4. Body mass index (BMI) <18.5 kg/m2 or >35 kg/m2
5. Burn injury
6. Any severe, persistent blood coagulation disorder with uncontrolled bleeding
7. Any congenital errors of amino acid metabolism
8. Uncontrolled hyperglycaemia despite insulin treatment
9. Known hypersensitivity to fish, egg, soybean proteins, peanut proteins, or to any of the active substances or excipients contained in SmofKabiven® extra Nitrogen or Olimel N9E
10. Known hypersensitivity to milk protein or to any other substance contained in Fresubin® Original
11. Treatment-refractory cardiopulmonary or metabolic instability showing persistent or progressive worsening despite increased interventions, including severe pulmonary oedema, severe cardiac insufficiency, myocardial infarction, acute phase of circulatory shock, severe sepsis, embolism, haemodynamic instability, metabolic or respiratory acidosis, hypotonic dehydration, or hyperosmolar coma
12. Severe renal dysfunction, defined as serum creatinine ≥2.0 times baseline or urine output <0.5 mL/kg/h for ≥12 hours (Acute Kidney Injury stage ≥2; [KDIGO 2012]), and blood urea nitrogen (BUN) exceeding 2 x upper limit of normal (ULN)
13. Severe liver failure with encephalopathy, including intoxication (e.g. paracetamol, death cap, golden chain) and/or liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma glutamyl transferase [GGT]) or bilirubin exceeding 5 x ULN
14. Oncologic disease with anticancer drug and/or radiation treatment incl. Hyperthermic Intraperitoneal Chemotherapy (HIPEC) during this Trial up to and including Study Day 28
15. Preceding transplantation causal for acute critical illness
16. Hemophagocytic syndrome
17. Pregnancy or lactation
18. Receiving end-of-life-care
19. Pathologically altered blood pH (arterial pH <7.0), oxygen saturation (SaO2 <80%), or carbon dioxide concentration (PaCO2 ≥80 mm Hg)
20. Hyperlipidaemia or any disorder of lipid metabolism characterised by hypertriglyceridaemia (serum triglyceride levels >4 mmol/L [>350 mg/dL])
21. Treatment-refractory, clinically significant major abnormality in the serum concentration of any electrolyte (sodium, potassium, magnesium, total calcium, chloride, inorganic phosphate)
22. Administration of growth hormone including teduglutide within the previous 4 weeks before randomisation
23. Invasive devices and procedures influencing metabolism and organ perfusion, e.g. extracorporeal membrane oxygenation (ECMO), continuous renal replacement therapy (CRRT), molecular absorbent recycling system (MARS), intra-aortic balloon pump (IABP)
24. Receipt of the last dose of study drug in another interventional clinical trial within the previous 4 weeks before randomisation into this clinical trial
25. Previous inclusion in the present study
26. Any other known reason that may prevent a patient to take part in the study in accordance with local requirements

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching ≥70% of the cumulative target for protein delivery from Study Day 2 through Study Day 6 | 5 days
  The cumulative target for protein delivery is 6.75 g/kg over 5 Study Days (based on a daily target of 0.75 g/kg/day on Study Day 2 and 1.5 g/kg/day on Study Days 3 through 6); 70% of the cumulative target for protein delivery is 4.73 g/kg.
  The cumulative protein delivery is calculated as the cumulative intake of amino acids from study drug and protein from enteral or oral nutrition on Study Day 2 through Study Day 6.

SECONDARY OUTCOMES:
Percentage of the cumulative target for protein delivery reached from Study Day 2 through Study Day 6 | 5 days
  Actual cumulative protein delivery (g/kg/5d) divided by 6.75 (g/kg/5d) and multiplied by 100.
Mean cumulative protein delivery by parenteral, enteral, and oral nutrition from Study Day 2 through Study Day 6 | 5 days
Calculated mean cumulative protein deficit during the period from Study Day 2 through Study Day 6 | 5 days
  The cumulative protein deficit is calculated as the cumulative target for protein delivery (6.75 g/kg/5d) minus the actual administered dose (g/kg/5d amino acids from study drug + g/kg/5d from enteral and oral nutrition.

OTHER OUTCOMES:
Mean total cumulative energy intake from parenteral, enteral and oral nutrition and from non-nutritional sources during the 5-day treatment period (calculated for each day from Study Day 2 through Study Day 6) | 5 days
Time to increase of daily enteral and oral nutrition intake above 20% of total energy target of 20 kcal/kg/d during the 5-day treatment period | 5 days
Mean daily insulin dose during the 5-day treatment period | 5 days
Mean cumulative insulin dose for the 5-day treatment period | 5 days
Mean change from baseline in daily insulin dose (Study Day 2 through Study Day 6) | 5 days
Maximum single insulin dose during the 5-day treatment period | 5 days
Mean maximum daily blood glucose value during the 5-day treatment period | 5 days
Mean minimum daily blood glucose value during the 5-day treatment period | 5 days
Mean blood glucose value during the 5-day treatment period | 5 days
Mean change from baseline in mean daily blood glucose value (Study Day 2 through Study Day 6) | 5 days
Change from baseline in SOFA score, calculated daily from Study Day 3 through Study Day 7 | 5 days
Overall survival time up to Study Day 28 | 28 days
All-cause mortality up to Study Day 28 | 28 days
Length of stay in the ICU up to Study Day 28 | 28 days
Re-admission to ICU up to Study Day 28 | 28 days
ICU mortality up to Study Day 28 | 28 days
Length of stay in the hospital up to Study Day 28 | 28 days
Re-admission to hospital up to Study Day 28 | 28 days
Hospital mortality up to Study Day 28 | 28 days
Therapeutic Intervention Scoring System (TISS)-28 score (including individual item score, category score, and total score) | Study Day 7
Duration of mechanical ventilation up to Study Day 28 | 28 days
Change from baseline of the Medical Research Council (MRC) sum score | Study Day 7, and either on day of ICU discharge or on Study Day 28, whatever occurs first
Change from baseline of ICU Mobility Scale | Study Days 7, 14, and 28
  Reference for ICU Mobility Scale: Hodgson C, Needham Dale, Haines K, Bailey M, Ward A, Harrold M, Young P, Zanni J, Buhr H, Higgins A, Presneill J, Berney S. Feasibility and inter-rater reliability of the ICU Mobility scale. Heart Lung 2014; 43(1):19-24. Erratum. Heart Lung 2014;43(4):388.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Bohe, Prof. MD, Principal Investigator — Département d'Anesthésie-Réanimation, Centre Hospitalier Lyon Sud, France
Locations (3):
- Hôpital Saint-Antoine, Département d'Anesthésie-Réanimation, Paris, France
- Klinikum rechts der Isar, Klinik für Anaesthesiologie, München, Germany
- SP ZOZ Wojewódzki Szpital Zespolony im. J. Śniadeckiego, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No